CLINICAL TRIAL: NCT05354297
Title: Evidence for Health Improvement in People With Diabetes Using One Touch & Partner Solutions (ECLIPSE)
Brief Title: Evidence for Health Improvement in People With Diabetes Using One Touch & Partner Solutions
Acronym: ECLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LifeScan (Industry)
Collaborators: Evidation Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062350
Record Dates: First submitted 2022-04-18; First posted 2022-04-29 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Cecelia Health (Experimental): Access to live Cecelia health coach on the telephone for 1 year plus access to Cecelia health coach by text messaging (via the OneTouch Reveal mobile diabetes app). Subjects will be provided with the OneTouch Verio Reflect glucose meter and the OneTouch Reveal (OTR) diabetes app.
  Interventions: Device: Cecelia Health plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app
- Fitbit (Experimental): Fitbit Inspire 2 wearable plus 1 year subscription to premium Fitbit application. Subjects will also be provided with the OneTouch Verio Reflect glucose meter and the OneTouch Reveal (OTR) mobile diabetes app.
  Interventions: Device: Fitbit plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app
- Noom (Experimental): Noom behavioural weight loss program subscription for 1 year. Subjects will also be provided with the OneTouch Verio Reflect glucose meter and the OneTouch Reveal (OTR) mobile diabetes app.
  Interventions: Device: Noom plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app
- Welldoc (Experimental): Multi-condition support program from Welldoc subscription for 1 year. Subjects will also be provided with the OneTouch Verio Reflect glucose meter.
  Interventions: Device: Welldoc plus OneTouch Verio Reflect® BGM and Welldoc app

INTERVENTIONS:
Device: Cecelia Health plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app — Expert guidance via coaching
  Arms: Cecelia Health
Device: Fitbit plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app — Fitness and wellness guidance
  Arms: Fitbit
Device: Noom plus OneTouch Verio Reflect® BGM and OneTouch Reveal® mobile app — Behavioral weight loss program
  Arms: Noom
Device: Welldoc plus OneTouch Verio Reflect® BGM and Welldoc app — Multi condition support
  Arms: Welldoc

SUMMARY:
ECLIPSE will evaluate the clinical and economic value of OneTouch Solutions in a real world study design. OneTouch Solutions describes a selection of devices and health and wellness solutions that people with diabetes (PWDs) can access online via OneTouch Solutions (Cecelia Health, Fitbit, Noom or Welldoc, each in combination with OneTouch Verio Reflect® blood glucose meter and the OneTouch Reveal® mobile app (or Welldoc app for the Welldoc arm)). ECLIPSE is a large parallel arm digital health study combining advanced blood glucose monitoring solutions with a choice of four different health and wellness applications or services. There are four unique study arms that will run in parallel over one year. The primary (A1c) endpoint for each study arm will be after 6 months and subjects will continue to use the interventions for a full year to generate data on sustained engagement with these products and services, and to collect healthcare utilization and health insurance claims information. Each study arm will differ to some degree in terms of patient baseline demographics (since subjects self-select their own app/intervention) and the experience per arm will be unique, and therefore each study arm will be analysed separately in terms of endpoints and outcomes.

DETAILED DESCRIPTION:
ECLIPSE (Evidence for health improvement in people with diabetes using One Touch & Partner Solutions) is a large parallel arm digital health study that will allow people with diabetes (PWDs) the freedom to choose the solution that is right for them, rather than forcibly randomize subjects to a specific study intervention. The intention of this real world study design is to mimic the choice PWDs will have when selecting a diabetes & digital health solution from the OneTouch Solutions website.

A target of 800 people with type 2 diabetes (PwT2Ds) will be recruited and offered one of four interventions with the aim of following 200 PWDs per study arm. Subjects in all four study arms will use a bluetooth connected OneTouch Verio Reflect blood glucose meter (BGM) which features a dynamic color range indicator (DCRI) and blood sugar mentor (BSM) insights. Subjects in three of the four study arms will also sync their Reflect BGM to the OneTouch Reveal (OTR) mobile diabetes app to enable further insights (PWDs in the Welldoc study arm will not use the OTR app).

The 4 unique study arms will also offer PWDs one of the following Partner offerings;

1. Cecelia Health, which offers guidance from certified Diabetes Care and Education Specialists
2. Fitbit, which offers activity and wellbeing insight from use of the Fitbit Inspire 2 tracker, and Fitbit Premium subscription
3. Noom, a psychology-based weight and wellness program
4. Welldoc, which offers personalized health coaching on multiple conditions, namely prediabetes, diabetes, hypertension and heart failure

ECLIPSE will gather glycemic measures, medication adherence, a variety of patient reported outcomes and partner app usage and app engagement analytics over one year. Health economic data (HECON) from PWDs from the year of participation in ECLIPSE will be analysed from a purchased dataset and a comparison will be made to HECON data from the same PWDs for the year prior to taking part in the study. In addition, a matched control group of PwT2D from the same purchased dataset will be compared to the data from all four study arms.

ELIGIBILITY:
Inclusion Criteria:

* Self reports a diagnosis of type 2 diabetes
* HbA1c ≥7.5% but ≤12% at screening
* Currently instructed by a health care provider (HCP) to use a blood glucose meter to test blood sugar
* Has a compatible smartphone and willing to redownload apps if they change phones during the study
* Has a stable and consistent home and/or office internet connection
* Currently on at least 1 oral (by mouth) or injected anti-diabetic medication (for lowering your blood glucose) with or without insulin therapy (insulin injections or an insulin pump) at screening

Exclusion Criteria:

* Currently pregnant or planning to be pregnant in the next 12 months
* Body Mass Index < 27
* Currently using a CGM (Continuous glucose monitor) or have used a personal CGM in the past 3 months
* Currently using a OneTouch Verio Reflect meter
* For FitBit arm only: Currently uses related fitness applications (e.g., MyFitnessPal, JEFIT, Fitness Coach, Yoga-Go, etc.) or wearable device (e.g., Fitbit, Apple Watch, Garmin, Withings, etc.) in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-07-26 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in A1c from screening to 3 and 6 months in each of the OneTouch Solutions programs | 3 and 6 months

SECONDARY OUTCOMES:
Change in mean blood glucose derived from blood glucose testing throughout the study in each of the OneTouch Solutions programs | 3 and 6 months
Change from baseline in diabetes distress as assessed by the diabetes distress scale (DDS) after 3 and 6 months | 3 and 6 months
Change from baseline in well-being as assessed by the WHO-5 survey after 3 and 6 months | 3 and 6 months
Change from baseline in patient activation measures as assessed by PAM-13 survey after 3 and 6 months | 3 and 6 months
Change from baseline in medication adherence as assessed by a medication adherence survey after 3 and 6 months | 3 and 6 months

OTHER OUTCOMES:
Changes over time in the number of app sessions performed within each of the OneTouch Solutions programs | Over 1 year
Change from baseline in A1c as a function of the number of app sessions performed within each of the OneTouch Solutions programs | Over 1 year
Quantify the number of medical insurance claims made by subjects within each of the OneTouch Solutions programs using data harvested from a large medical insurance dataset | Over 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Nchih Lee, PhD, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No